CLINICAL TRIAL: NCT02711618
Title: Clinical Study to Evaluate the Performance of the UltraShape Contour I V3 for Non-Invasive Abdominal Fat Reduction Among Patients With BMI Above 28
Brief Title: Non-Invasive Abdominal Fat Reduction With BMI Above 28
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF19571
Record Dates: First submitted 2016-02-25; First posted 2016-03-17 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Unwanted Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UltraShape Contour I V3 treatment (Experimental): Up to 60 healthy adult volunteers seeking noninvasive fat reduction, male and females at up to four sites, age of 18 to 60, with BMI above 28
  Interventions: Device: UltraShape Contour I V3

INTERVENTIONS:
Device: UltraShape Contour I V3 — Tissue selectivity is achieved by a proprietary knowledge of parameters ensuring specific destruction of the fat cells only within the target area. All other types of tissue, such as blood vessels, muscles and peripheral nerves remain intact. There are no thermal effects. Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time
  Other Names: Contour I V3

SUMMARY:
Prospective, one arm, baseline-controlled clinical study for the evaluation of UltraShape contour I V3 for non-invasive fat reduction.

The study will conduct using the UltraShape contour I V3 using U-Sculpt/VDF transducer on the abdomen.

DETAILED DESCRIPTION:
This study is a prospective, one arm, up to four sites, clinical study showing the performance and safety of the UltraShape contour I V3 device non-invasive abdominal fat reduction for subjects with body mass index (BMI) above 28.

Up to 60 healthy subjects will be enrolled. All subjects will undergo an assessment of their general health. During the treatment period, subject's fat thickness and circumferences will be measured and three successive UltraShape contour I V3 treatments will be performed (two weeks interval).

Subjects will undergo treatment with the UltraShape contour I V3 using the U-Sculpt/VDF transducer on the abdomen area.

Follow-up (FU) visits will be conducted as follows: 4 weeks FU, 8 weeks FU and 12 weeks FU post last treatment (Tx.3). Subject's fat thickness and circumference will be measured at each visit. Subject's blood test will be taken at baseline (prior to the first treatment, pre Tx.1), before the third treatment (pre Tx.3) and at 12 weeks follow-up visit (12wk FU). "No Pregnancy" will be verified before first treatment as well. In all following visits (TX2, Tx3 and FU 1 FU 2 and FU3), lack of pregnancy will be verified by questioning. Additionally, subject satisfaction and investigator satisfaction questionnaires will be completed at each FU visit. Finally, photography will be performed under visible light conditions of the front, right and left view. Optional, 3D photographs will be taken at each visit (at treatment visits, prior to treatments).

ELIGIBILITY:
Inclusion Criteria:

subject is eligible to participate in the study if he or she meets all the following inclusion criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects,18 and 60 years of age at the time of enrolment
3. Fitzpatrick Skin Type I to VI.
4. Abdominal fat thickness of at least 1.5 cm (measured by calibrated caliper).
5. BMI above 28 (normal to overweight).
6. If female, not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e. oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. Negative urine pregnancy test as tested before the first treatment for women with bearing potential (e.g. not menopause). In addition, negative pregnancy following pregnancy inquiry for each visit (treatments and follow up), starting from the second treatment.
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations

Exclusion Criteria:

A subject is not eligible for participation in this study if he/she meets any of the following exclusion criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Current hyperlipidemia, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease or malignancy
3. Previous liposuction or body contouring procedures in the treatment areas of the abdomen or flanks. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing.
4. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area.
5. Poor skin quality (i.e., laxity).
6. Abdominal wall diastasis or hernia on physical examination.
7. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months.
8. Childbirth within the last 12 months or breastfeeding women.
9. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study.
10. Unstable weight within the last 6 months (i.e., ± 3 percent weight change in the prior six months).
11. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
12. Abdominal fat thickness lower than 2.5 cm after strapping.
13. Participation in another clinical study within the last 6 months.
14. Non-invasive body-contouring procedures in the treatment area completed less than twelve months prior to study enrollment.
15. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change in abdominal fat thickness compared to baseline | Baseline and 12 weeks
  Abdominal fat thickness reduction post UltraShape contour I V3 treatments at 12 weeks follow-up (12wk FU) versus baseline.

SECONDARY OUTCOMES:
Change in abdominal fat thickness compared to baseline | Baseline, 8 weeks and 16 weeks
  Abdominal fat thickness reduction as measured by Ultrasound device post UltraShape contour I V3 treatments at follow-up visits
Change in abdominal fat thickness compared to baseline | Baseline, 8 weeks, 12 weeks, and 16 weeks
  Abdominal fat thickness reduction as measured by caliper post UltraShape contour I V3 treatments at follow-up visits versus baseline
Change in abdominal circumference reduction compared to baseline | Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  Abdominal circumference reduction post UltraShape contour I V3 treatments at all treatment visits and follow-up visits
Blood panel and fat lipid profile compared to baseline levels | Baseline, 4 weeks and 16 weeks
  Blood elements levels (e.g. lipids, Glucose) before the third treatment (at 4 weeks) and at the last follow-up visit (at 16 weeks) versus baseline
Investigator satisfaction | 8 weeks, 12 weeks, and 16 weeks
  Investigator satisfaction: success is defined as when at least 50% of the observations are ranked as at least satisfied by the study investigator at each of the follow up visits
Subject satisfaction | 8 weeks, 12 weeks, and 16 weeks
  Subject satisfaction: success is defined as when at least 50% of the subjects are satisfied with treatment results at each of the follow up visits
Comfort level during treatment | day 0, 2 weeks, and 4 weeks
  Comfort assessment will be performed independently by subjects using a numerical scale. Subjects will assess treatment comfort immediately post each of the three treatments

OTHER OUTCOMES:
Number of participants with adverse events | day 0 until 16 weeks
  Description, severity, intervention and outcome of adverse events will be reported on an adverse event form and number of participants will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Gold, M.D., Principal Investigator — Aesthetic Plastic Surgery & Cosmetic Medicine Great Neck, New York
Locations (3):
- United States (3):
  - Sanctuary Plastic Surgery, Boca Raton, Florida
  - 833 Northern Boulevard, Great Neck, New York
  - Laser and Skin Surgery Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arner P. Regional adipocity in man. J Endocrinol. 1997 Nov;155(2):191-2. doi: 10.1677/joe.0.1550191. No abstract available. PMID 9415044